CLINICAL TRIAL: NCT01391156
Title: Efficacy of 3% Minoxidil Versus Combined 3% Minoxidil and 0.1% Finasteride for Male Pattern Hair Loss: a Randomized, Double-blinded, Comparative Study
Brief Title: Efficacy Study of Minoxidil Lotion Versus Combined Minoxidil and Finasteride Lotion to Treat Male Pattern Hair Loss
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mae Fah Luang University Hospital (Other)
Responsible Party: Principal Investigator, Chuchai TANGLERTSAMPAN, MD, Chuchai Tanglertsampan, MD, Mae Fah Luang University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: REH-54015
Record Dates: First submitted 2011-07-01; First posted 2011-07-11 (Estimated); Last update posted 2012-07-20 (Estimated); Status verified 2012-07

CONDITIONS: Androgenetic Alopecia
Keywords: minoxidil; finasteride; topical; lotion; male pattern hair loss; androgenetic alopecia
MeSH Terms: conditions — Alopecia | interventions — Minoxidil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Minoxidil (Experimental)
  Interventions: Drug: 3%Minoxidil lotion
- MinoxidilFinasteride (Active Comparator)
  Interventions: Drug: 3% Minoxidil with 0.1% Finasteride lotion

INTERVENTIONS:
Drug: 3%Minoxidil lotion — 3% Minoxidil lotion apply two times a day
  Arms: Minoxidil
Drug: 3% Minoxidil with 0.1% Finasteride lotion — 3% Minoxidil with 0.1% Finasteride lotion apply two times a day.
  Arms: MinoxidilFinasteride

SUMMARY:
The purpose of this study is to compare the efficacy of 3% Minoxidil lotion and 3% Minoxidil with 0.1% Finasteride lotion for 6 months in male pattern hair loss.

ELIGIBILITY:
Inclusion Criteria:

* male, age 18-15 years
* androgenetic alopecia grade 3V to 5 ( Norwood-Hamilton classification)

Exclusion Criteria:

* use minoxidil in 6 months
* use finasteride in 12 months
* use ketoconazole, tar, selenium shampoo, topical tretinoin, topical steroid in 2 weeks
* seborrheic dermatitis or psoriasis on scalp
* history of allergy to minoxidil, finasteride

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2011-03; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
The mean change of hair count from baseline and 6 months | baseline and 6 months
  Total hair count on the vertex is measured on 1 cm2 circular area. The mean change in hair count is compared at baseline and 6 months.The significance of change is determined by Unpaired t Test.

SECONDARY OUTCOMES:
Global photographic assessment by dermatologists | baseline and 6 months
  Photographs of the vertex scalp are taken at baseline and 6 months. A panel of 3 dermatologists assesssed the change in hair growth using a 7-point scale.

CONTACTS AND LOCATIONS:
Overall Officials: Chuchai Tanglertsampan, MD, Principal Investigator — Mae Fah Luang University Hospital(Bangkok)
Locations (1):
- Mae Fah Luang University Hospital(Bangkok), Bangkok, Bangkok, Thailand